CLINICAL TRIAL: NCT06036212
Title: A Prospective, Single-blind, Multi-Centre, Randomised Controlled Study to Evaluate the Clinical and Patient Reported Outcomes Following Unicompartmental Knee Arthroplasty With a Robotic Assisted Technique
Brief Title: Study to Evaluate Patient Outcomes and Safety and Effectiveness of Robotic Assisted Unicompartmental Knee Replacements Versus Conventional Unicompartmental Knee for Subjects With Primary Arthritis of the Knee Joint Involving One (UKA) Compartment (Medial or Lateral)
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Terminated post suspension, no subjects enrolled
Sponsor: Smith & Nephew, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2022.03 Robotics JII UK RCT
Record Dates: First submitted 2023-09-06; First posted 2023-09-13 (Actual); Last update posted 2025-11-17 (Actual); Status verified 2025-10

CONDITIONS: Arthroplasty, Replacement, Knee; Unicompartmental Knee Arthroplasty
Keywords: Robotics assisted surgery; Computer assisted surgery; Unicompartmental knee arthroplasty; Unicompartmental knee replacement; Partial knee replacement; Partial knee arthroplasty; Journey II UK

STUDY DESIGN:
Who Masked: Participant
Masking Description: Single-blinded to study participant. The study participants will not be aware of the treatment received. For those not being put under general anesthetic during the procedure, a screen will be put up between the subjects face and the ongoing procedure and associated platforms/instrumentation so that they are unable to see any of the procedure and are unable to guess whether they are having robotics assisted surgery or conventional surgery. Extra incisions (maximum of 4 based on approach that the operating surgeon uses) are required to conduct robotic assisted surgery, those subjects receiving conventional surgery will receive sham incisions.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Journey II UK Partial Knee Implant with Robotic Assisted Surgery (Experimental): Robotically-assisted implant of the partial (unicompartmental) knee implant (Journey II UK)
  Interventions: Device: Robotic System
- Journey II UK Partial Knee Implant with Conventional, Manual Surgery (Sham Comparator): Implant of the partial (unicompartmental) knee implant (Journey II UK) with conventional, typical manual surgery
  Interventions: Device: Conventional

INTERVENTIONS:
Device: Robotic System — Robotic assisted Unicompartmental Knee replacement (UKA)
  Arms: Journey II UK Partial Knee Implant with Robotic Assisted Surgery
Device: Conventional — Unicompartmental Knee Arthroplasty (UKA) with conventional approach and conventional manual instrumentation
  Arms: Journey II UK Partial Knee Implant with Conventional, Manual Surgery

SUMMARY:
The overall aim of this trial is to compare functional and patient-reported outcomes and to assess the safety and effectiveness and long-term performance of the Smith+Nephew Robotic Systems for Unicompartmental Knee Replacements to non-robotic, conventionally implanted Unicompartmental Knee Replacements.

DETAILED DESCRIPTION:
There are two phases for this study:

* Phase 1: The primary objective of this study is to compare Forgotten Joint Score (FJS) 12-month patient reported outcome scores, in patients undergoing robotic assisted Unicompartmental Knee Replacements as compared to those undergoing conventionally implanted Unicompartmental Knee Replacements
* Phase 2: The primary objective of Phase 2 of this study is evaluate the revisions rates of the JII UK unicompartmental knee at 10 years

Research participants / locations:

280 research participants will be recruited from up to 15 sites in the UK, US and Europe. There will be 140 participants undergoing robotic assisted Unicompartmental Knee Replacements and 140 participants undergoing non-robotic, conventionally implanted Unicompartmental Knee Replacements.

ELIGIBILITY:
Inclusion Criteria:

1. The subject or, legal guardian (in the case of difficulty reading and/or writing,) must provide written informed consent, including consent for any incidental findings to be reported to their General Practitioner (reference section 7.5).
2. Subjects eighteen (18) years and older and considered to be skeletally mature at the time of surgery.
3. Willing and able to make all required study visits (for both phases of the study, up to 10 years postoperatively).
4. Able to follow instructions and deemed capable of completing all the study questionnaires.
5. The subject has primary arthritis of the knee joint involving one (UKA) compartment (medial or lateral), and is suitable for JOURNEY II UK in the opinion of the surgeon.
6. The subject can, and is willing to have radiographic images taken to include non-standard of care imaging (for long leg radiographs at follow up).

Exclusion Criteria:

1. Contraindications or hypersensitivity to the use of the JII UK implant components (e.g., oxinium femoral, Tibial Baseplate, XPLE insert).
2. The subject is contraindicated for the use of robotic-assisted knee arthroplasty.
3. Participation in the treatment period of another clinical trial within thirty (30) days of the preoperative visit, or during the study.
4. Women who are pregnant, nursing, or of child-bearing potential who are not utilizing highly effective birth control measures.
5. Any subject that meets the definition of a Vulnerable Subject per ISO 14155 Section 3.55.
6. Subjects who have participated previously in this trial through UKR on other knee.
7. The subject is listed for a simultaneous bilateral knee arthroplasty
8. Subjects experiencing severe pain in both knees and consequently anticipating bilateral surgery within 12 months.
9. The subject requires a complex implant or any other implant, other than a standard UKR (e.g. stems, augments or custom-made devices)
10. Subject has an active infection or sepsis or has had previous intra-articular infections
11. Subjects with a history of poor compliance with medical treatment
12. The subject, in the opinion of the investigator, has a neuromuscular disorder (e.g. Charcot joint) that prohibits control of the index joint
13. Cases where bone stock is poor and would therefore make the procedure unjustifiable
14. Subjects with a BMI of 40 or higher
15. Those with incomplete/sufficient soft tissue around the joint.
16. Subjects with Conditions that tend to place increased loads on implants such as age, weight, and activity level, which are incompatible with a satisfactory long-term result.
17. Subjects with a medical or physical condition that, in the opinion of the Investigator, would preclude safe subject participation in the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2023-11-21 (Actual); Primary Completion 2027-03-15 (Estimated); Study Completion 2036-03-15 (Estimated)

PRIMARY OUTCOMES:
Forgotten Joint Score 12 (FJS-12) at 12 Months Post Operative | 12 months post operative
  The Forgotten Joint Score 12 (FJS-12) is a self-administered score where subjects are asked to rate their awareness of their knee arthroplasty in 12 questions with a five-point Likert response format: "Never", "almost never", "seldom", "sometimes" and "mostly". The item scores are summed and linearly transformed in a 0 to 100 scale with a high value reflecting the ability of the subject to forget about the replaced knee joint during the activities of daily living.
Implant Survival at 10 years | 10 years post operative
  Number of participants with implant survival at 10 years with survival defined as lack of unicompartmental knee arthroplasty (UKA) revision.

SECONDARY OUTCOMES:
Oxford Knee Score (OKS) | Pre-operative, 6 weeks, 6 months, 1 year, 2 years, 5 years, 10 years post operative
  The Oxford Knee Score (OKS) is a self-administered score contains 12 equally weighted questions on activities of daily living. Responses to each question range from 0-4 with a range of a possible overall score from 0-48. A score of 0 is the worst possible outcome while a score of 48 is the best possible outcome.
Oxford Arthroplasty Early Recovery Score (OARS) | Day 1, day 2, day 3, day 7, day 14, 6 weeks post operative
  The Oxford Arthroplasty Early Recovery Score (OARS) is a self-administered score regarding how the participant is feeling consisting of four domains: Pain, Sleep, Nausea and feeling unwell, and Mobility. The OARS questionnaire is scored 0-100 with zero being a poor recovery and 100 being positive and indicative of a good recovery.
Oxford Arthroplasty Early Change Score (OACS) | Day 1, day 2, day 3, day 7, day 14, 6 weeks post operative
  The Oxford Arthroplasty Early Change Score (OACS) is a self-administered score regarding how the participant feels after their surgery, compared to before, concentrating on areas such as ability, pain, overall feelings. The OACS questionnaire is scored from negative 50 to positive 50 with minus 50 being much worse than before surgery to 50 being much better than before surgery. Zero indicates no change from self-reported pre-operative health status.
EuroQol Five-Dimensional Five-Level (EQ-5D-5L) - Descriptive System | Pre-operative, 6 weeks, 6 months, 12 months, 2 years, 5 years, 10 years post operative
  The descriptive system is used to describe the subject's health state & consists of 5 dimensions: mobility, self-care, usual activities, pain/discomfort, and anxiety/depression. Each dimension has 5 levels to choose the most appropriate answer: no problems, slight problems, moderate problems, severe problems, and extreme problems. The subject is asked to indicate his/her health state by marking the most appropriate statement in each of the five areas. Responses are coded as single-digit numbers expressing the severity level selected in each dimension. For instance, 'slight problems' (e.g. 'I have slight problems in walking about') is always coded as '2'. The digits for the 5 dimensions are combined in a 5-digit code. The EQ- 5D-5L index value is derived by using the vendor supplied calculator to convert each 5-digit EQ-5D-5L profile. A higher number is a better outcome.
EuroQol Five-Dimensional Five-Level (EQ-5D-5L) - Visual Analogue Scale (VAS) | Pre-operative, 6 weeks, 6 months, 12 months, 2 years, 5 years, 10 years post operative
  The EQ VAS records the subject's self-rated health on a vertical visual analogue scale. The endpoints on the scale are labelled "The best health you can imagine" and "The worst health you can imagine". Participants indicate a numerical value from 1-100 where 0 is the worst imaginable health state and 100 is the best imaginable health state. The VAS can be used as a quantitative measure of health outcome as judged by the individual respondents.
Visual Analogue Scale (VAS) - Pain Score | Pre-operative, 6 weeks, 6 months, 12 months, 2 years, 5 years, 10 years post operative
  The Visual Analogue Score (VAS) - Pain Score is self-administered score assessing participant pain using Visual Analog Scale (VAS) assessments. Subjects will be asked to complete their pain levels on a scale of 0-100, 0 being no pain experienced and 100 meaning the worst pain possible.
Knee Injury and Osteoarthritis Outcome Score (KOOS) | Pre-operative, 12 months, 2 years, 5 years, 10 years post operative
  There are five patient-relevant subscales of the KOOS, and each are scored separately: Pain (9 items), Activities of Daily Living (ADL) function (17 items), Sport and Recreation Function (5 items), Symptoms (7 items), and Quality of Life (4 items).
  A Likert scale is used, and all items have five possible answer options scored from 0 (no problems) to 4 (extreme problems). Each of the 5 scores is calculated as the sum of the items included and then each score is transformed to a 0-100 scale, with 0 representing extreme knee problems and 100 representing no knee problems. An aggregate score is not calculated so that each of the 5 dimensions can be assess separately.
Implant Survival at 2 Years and 5 Years | 2 years and 5 years post operative
  Number of participants with implant survival at 2 years and 5 years with survival defined as lack of unicompartmental knee arthroplasty (UKA) revision.
Forgotten Joint Score 12 (FJS-12) | Baseline, 6 weeks, 6 months, 2 years, 5 years, 10 years post operative
  The Forgotten Joint Score 12 (FJS-12) is a self-administered score where subjects are asked to rate their awareness of their knee arthroplasty in 12 questions with a five-point Likert response format: "Never", "almost never", "seldom", "sometimes" and "mostly". The item scores are summed and linearly transformed in a 0 to 100 scale with a high value reflecting the ability of the subject to forget about the replaced knee joint during the activities of daily living.

CONTACTS AND LOCATIONS:
Overall Officials: Patricia McCracken, Study Director — Smith & Nephew, Inc.
Locations (5):
- United Kingdom (5):
  - The Royal Orthopaedic Hospital NHS Foundation Trust, Birmingham, West Midlands
  - Colchester General Hospital, Colchester
  - Central Middlesex Hospital, London
  - Imperial College Healthcare NHS Trust, St Mary's Hospital, London
  - Norfolk and Norwich University Hospital NHS Foundation Trust, Norwich

IPD SHARING:
Plan to Share IPD: No